CLINICAL TRIAL: NCT05863728
Title: Post-Operative Evaluation of Endodontic Microsurgeries Done Using a Piezoelectric Ultrasonic Technique: An in Vivo Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud Yehia Abouel Naga, Principal Investigator/ Assistant Lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31/5/2020
Record Dates: First submitted 2023-04-06; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Periapical Diseases; Endodontic Overfill; Healing Surgical Wounds
Keywords: Endodontic Microsurgery; Piezosurgery; Trephine bur
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezosurgery assisted group (Experimental): A Piezosurgery assisted cavity preparation was performed using a IM4A Piezosurgery tip mounted in the handpiece of a Piezosurgery device (PIEZOSURGERY touch, Mectron, Carasco, Italy) at an operating frequency in the range of 24 to 36 kHz with power ratings 55 W for osteotomy and root-end resection
  Interventions: Procedure: Piezosurgery assisted group
- Trephine Burs assisted group (Experimental): Trephine bur assisted cavity preparation was performed using a TPB-4 trephine bur mounted in 20:1 contra angled handpiece of an implant motor (ImplaNX, Micro-NX, Republic of Korea) at an operating speed in the range of 800 to 1200 / Torque 30 N for osteotomy and root-end resection
  Interventions: Procedure: Trephine Bur assisted group

INTERVENTIONS:
Procedure: Piezosurgery assisted group — apicectomy will be done using the Piezosurgery device
  Arms: Piezosurgery assisted group
Procedure: Trephine Bur assisted group — apicectomy will be done using the trephine burs
  Arms: Trephine Burs assisted group

SUMMARY:
The aim of the study was to evaluate the effect of Piezosurgery and Trephine bur as cutting tools on post-operative sequelae including pain and swelling following guided endodontic microsurgeries.

DETAILED DESCRIPTION:
Materials and Methods: Twenty healthy male patients aged between 18 and 45 years old were selected in the study. Mandibular first molar teeth with failed non-surgical treatment or re-treatment due to iatrogenic errors at the apical 3mm of the mesial root canal including canal ledging, zipping and transportation, root perforation, separated instrument, and canal calcification were selected. Piezosurgery assisted cavity preparation and root-end resection were performed in Groups I and II, and Trephine bur assisted cavity and root-end resection was performed in Groups III and IV. An apical curettage was performed and the over-extended objects such as separated instruments or gutta percha were removed. The PRF clots was placed inside the bone cavity in groups I and III while the bone cavity was kept for 2 min to allow the blood clots to be formed in groups II and IV. The degree of pain and swelling were recorded for five days every 24, 48, 72, 96, and 120 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Mandibular first molar teeth were selected according to specific inclusion criteria including:

1. Teeth presented with failed non-surgical treatment or re-treatment. Failure is due to iatrogenic errors at the apical 3mm of the mesial root canal including canal ledging, zipping and transportation, root perforation, separated instrument and canal calcification.
2. Teeth presented with normal pocket depth ranges from 1 to 3mm, up to grade II tooth mobility.
3. Teeth presented without periapical radiolucency (Class A) or with periapical radiolucency not more than 1 mm in diameter both mesiodistally and buccolingually (Class B) according to the preoperative endodontic microsurgical classification of teeth.
4. Teeth presented with non-fused mesial and distal roots and the mesial roots are range from 10 to 15 mm. in length, Type III root canal configuration (Two canals run separately from orifice to apex). The root canal curvature angle was measured using the Weine technique to be not less than 160° in both directions buccolingually and mesiodistally.
5. At the apical 3 mm of the mesial radiographic root apex, the distance from the outer surface of the buccal cortical plate of bone to the buccal side of the mesial root is 1.5 mm (Depth I). The buccolingual dimension of the mesial root is 7 mm mm (Depth II). The distance from the lingual surface of the mesial root to the outer surface of the lingual cortical plate of bone is 3.5 mm. (Depth III).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessment | 24 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative pain assessment | 48 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative pain assessment | 72 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative pain assessment | 96 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative pain assessment | 120 hours
  The postoperative pain assessment was done using the modified verbal descriptor scale as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).

SECONDARY OUTCOMES:
Postoperative swelling assessment | 24 hours
  Patients were instructed to the description of each level of swelling as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative swelling assessment | 48 hours
  Patients were instructed to the description of each level of swelling as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative swelling assessment | 72 hours
  Patients were instructed to the description of each level of swelling as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative swelling assessment | 96 hours
  Patients were instructed to the description of each level of swelling as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).
Postoperative swelling assessment | 120 hours
  Patients were instructed to the description of each level of swelling as follows; None (Score 0), Mild (Score 1), Moderate (Score 2), and Severe (Score 3).

OTHER OUTCOMES:
Post-operative CBCT scans | 6 months
  Evaluation of surgical endodontic healing according to Modified PENN 3D criteria
Post-operative CBCT scans | 12 months
  Evaluation of surgical endodontic healing according to Modified PENN 3D criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Cairo, Egypt